CLINICAL TRIAL: NCT05836454
Title: The Effect of Progressive Muscle Relaxation Technique and Myofascial Release Technique on Premenstrual Symptoms, Blood Circulation, and Quality of Life in Women With Premenstrual Syndrome: a Single-blind Randomized Controlled Study
Brief Title: The Soft Tissue Mobilization Techniques on PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMSBloodFlow
Record Dates: First submitted 2023-03-14; First posted 2023-05-01 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-05

CONDITIONS: Premenstrual Syndrome; Premenstrual Pain; Chronic Pelvic Pain
Keywords: myofascial releasing technique; progressive relaxation technique; blood flow velocity
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Intervention Model Description: Single Blind Randomized Controlled Study
Who Masked: Outcomes Assessor
Masking Description: Evaluations will be made by another physical therapist who is blinded to the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Progressive Muscle Relaxation Group: (Experimental): Progressive Muscle Relaxation technique will be applied to this group. Technique will be applied 3 days a week for 2 menstrual cycles.
  Interventions: Other: Progressive Muscle Relaxation Group:
- Myofascial Release Technique Group (Experimental): Myofascial Release Technique will be applied to this group. Technique will be applied 3 days a week for 2 menstrual cycles.
  Interventions: Other: Myofascial Release Technique Group
- Control Group (No Intervention): The control group will be asked to continue their normal lives.

INTERVENTIONS:
Other: Progressive Muscle Relaxation Group: — Progressive muscle relaxation is a relaxation technique that involves regular and sequential contraction and relaxation of muscles until the whole body is relaxed.
  Arms: Progressive Muscle Relaxation Group:
Other: Myofascial Release Technique Group — It is a physiotherapy technique based on soft tissue mobilization. All enveloping fascia sale prices are positive for mobility, a user used for adhesions and pain.
  Arms: Myofascial Release Technique Group

SUMMARY:
The aim of this study is investigate the effects of progressive relaxation and myofascial release technique on blood flow velocity, pain, premenstrual symptoms and quality of life in premenstrual syndrome patients. There are tree groups in the study. These groups are; progressive muscle relaxation group, myofascial relaxation technique and control group. Evaluations will be made by another physical therapist who is blinded to the groups. Participants will be evaluated within the first 3 days of their menstrual cycle. Baseline assessment and post- treatment assessment will be done. Follow-up evaluation will be done on the fifth cycle, two cycles after the post-treatment evaluation.

DETAILED DESCRIPTION:
The aim of this study is investigate the effects of progressive relaxation and myofascial release technique on blood flow velocity, pain, premenstrual symptoms and quality of life in premenstrual syndrome patients. The study planned as a single-blind randomized controlled trial. The volunteers who were invited to the study and signed the voluntary consent form will be randomized via random allocation software to divided into 3 groups. These groups are; progressive muscle relaxation group, myofascial relaxation technique and control group. Evaluations will be made by another physical therapist who is blinded to the groups. Participants will be evaluated within the first 3 days of their menstrual cycle. Baseline assessment will be done in the first 3 days of the first cycle, after first treatment acute assessment will be done. Post-treatment evaluation will be done in the first 3 days of the 3rd cycle after treatment for two cycles. Follow-up evaluation will be done in the first 3 days of the fifth cycle, two cycles after the post-treatment evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Pain score of 4 cm or more according to the Visual Analogue Scale.
* Having a regular menstrual cycle for 12 months (24-35 days).
* According to the International Physical Activity Questionnaire-Short Form (IPAQ-SF), the weekly Metabolic Equivalent of Task (MET) value is below 600 MET-min/week.

Exclusion Criteria:

* Those who have undergone surgery in the last 6 months,
* Those who use cigarettes and alcohol,
* Those who are pregnant,
* Those with urinary, genital, gastrointestinal disorders,
* Those who have had hysterectomy surgery will be excluded.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Blood Flow Rate at Two Menstrual Cycle | Baseline and 8 weeks
  Blood flow rate will be evaluated with the portable vascular doppler. Measurements will be made from the right or left common iliac artery, branches of the abdominal aorta, and the ipsilateral femoral artery. After the ultrasound gel is applied to the measurement area, the probe will be placed at an angle of 30° and the measurement will be taken.
Follow- up Evaluation Blood Flow Rate | 8 weeks through study completion
  Blood flow rate will be evaluated with the portable vascular doppler. Measurements will be made from the right or left common iliac artery, branches of the abdominal aorta, and the ipsilateral femoral artery. After the ultrasound gel is applied to the measurement area, the probe will be placed at an angle of 30° and the measurement will be taken.

SECONDARY OUTCOMES:
Change from Baseline Pain Severity at Two Menstrual Cycle | Baseline and 8 weeks
  It will be evaluated with the visual analog scale. Pain is determined by measuring the mark on the 10-centimeter line according to the severity of the pain. According to the Visual Analogue Scale (VAS), a score of 0 indicates no pain, and 10 indicates unbearable pain.
Follow-up Evaluation Pain Severity at Two Menstrual Cycle | 8 weeks through study completion
  It will be evaluated with the visual analog scale. Pain is determined by measuring the mark on the 10-centimeter line according to the severity of the pain. According to the VAS, a score of 0 indicates no pain, and 10 indicates unbearable pain.
Change from Baseline Pain Threshold at Two Menstrual Cycle | Baseline and 8 weeks
  It will be evaluated with a digital algometer and the value on the algometer will be recorded in kg. Evaluation areas are Vastus medialis, Pectoralis major, Gluteus maximus, Gluteus medius, Iliopsoas, Lumbal paraspinal, Trapezius, Spina iliaca anterior superior (SIAS). Measurements will be made from the muscle body.
Follow-up Evaluation Pain Threshold | 8 weeks through study completion
  It will be evaluated with a digital algometer and the value on the algometer will be recorded in kg. Evaluation areas are Vastus medialis, Pectoralis major, Gluteus maximus, Gluteus medius, Iliopsoas, Lumbal paraspinal, Trapezius, Spina iliaca anterior superior (SIAS). Measurements will be made from the muscle body.
Change from Baseline Premenstrual Syndrome at Two Menstrual Cycle | Baseline and 8 weeks
  It will be evaluated with the premenstrual symptom scale. Evaluates the symptoms related to premenstrual syndrome in detail.
Follow-up Evaluation Premenstrual Syndrome | 8 weeks through study completion
  It will be evaluated with the premenstrual symptom scale. Evaluates the symptoms related to premenstrual syndrome in detail.
Change From Baseline Health-related Quality of Life at Two Menstrual Cycle | Baseline and 8 weeks
  It will be evaluated with the SF-36 short form. Turkish validity and reliability study made by Kocyigit et al. In the evaluation of the scale, a score between 0-100 points can obtained from each sub-dimension, 0 points indicates that the quality of life dimension is bad and 100 points that it is good.
Follow-up Evaluation Health-related Quality of Life | 8 weeks through study completion
  It will be evaluated with the SF-36 short form. Turkish validity and reliability study made by Kocyigit et al. In the evaluation of the scale, a score between 0-100 points can obtained from each sub-dimension, 0 points indicates that the quality of life dimension is bad and 100 points that it is good.

CONTACTS AND LOCATIONS:
Overall Officials: Çisel Demiralp, Msc, Principal Investigator — Eastern Meditteranean Univeristy
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided